CLINICAL TRIAL: NCT04031443
Title: The Prescription Pattern and Awareness About Antibiotic Prophylaxis and Resistance Among Pediatric Dentists (Cross Sectional Study)
Brief Title: Prescription Pattern and Awareness About Antibiotic Prophylaxis and Resistance
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa aly fouad elchaghaby, Lecturer of Pediatric Dentistry and Dental public health, Faculty of Dentistry, Cairo University, Egypt., Cairo University
Other Study IDs: antibiotic prescription
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Antibiotic Prescription
Keywords: prescription pattern; antibiotic prophylaxis; antibiotic resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the knowledge of Pediatric dentists regarding the prescription of antibiotics, antibiotic prophylaxis and antibiotic resistance

DETAILED DESCRIPTION:
Antibiotics commonly are prescribed by dentists, and the uses and abuses of these drugs should be familiar to all practicing clinicians. Antibiotics are used in dentistry for two major reasons: to control oral infection, and to prevent a bacteremia precipitated by dental manipulations from causing severe systemic sequelae.

In recent years, there has been an increasing tendency to reduce the widespread use of antibiotics for prophylactic and therapeutic purposes. This is based, both on increasing scientific evidence and enhanced professional experience. The development of resistant strains of microorganisms, doubt on the efficacy of the proposed prophylactic regimens, possible toxic and adverse reactions to antibiotics and poor compliance by patients and dentists raised questions about risks and benefits.

The American Academy of Pediatric Dentistry (AAPD) has published guidelines for antibiotic use, recognizing the increasing prevalence of antibiotic-resistant microorganisms. The guidelines are intended to provide guidance for the proper and judicious use of antibiotic therapy in the treatment of oral conditions in children.

Good knowledge about the indications of antibiotics is the need of the hour in prescribing antibiotics for dental conditions. Dental practitioners should know the protocol to be applied in their patients and should apply the most recent guidelines regarding antibiotic regimen.

ELIGIBILITY:
* Inclusion criteria:

  * Dental practitioner
  * Deal with children
* Exclusion criteria:

  * Undergraduate student

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: dental practitioner who deal with children
Sampling Method: Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
The prescription pattern of antibiotics among Pediatric dentists | 1 month
  measured by Questionnaire and the measuring unit is binary yes or no

SECONDARY OUTCOMES:
Most common antibiotic prescribed, duration and dosage | 1 month
  measured by Questionnaire and the measuring unit is open ended questions
Clinical conditions for which antibiotics were prescribed | 1 months
  measured by Questionnaire and the measuring unit is Multiple choice questions
Awareness about antibiotic prophylaxis | 1 month
  measured by Questionnaire and the measuring unit is binary yes or no
Awareness about antibiotic resistance | 1 month
  measured by Questionnaire and the measuring unit is binary yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt